CLINICAL TRIAL: NCT07173803
Title: The Progressive Supranuclear Palsy Clinical Trial Platform
Acronym: PTP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adam Boxer (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Alzheimer's Therapeutic Research Institute (Other); University of Southern California (Other); Massachusetts General Hospital (Other); University of California, San Diego (Other); Alzheimer's Clinical Trials Consortium (Other)
Responsible Party: Sponsor-Investigator, Adam Boxer, Endowed Professor in Memory and Aging, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATRI-015; R01AG085029 (NIH)
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Progressive Supranuclear Palsy(PSP)
Keywords: PSP; Placebo-Controlled; Double-Blind; Master Protocol
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — AADvac1; LM11A-31

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A: AADvac1 (Experimental): Participants are randomized to receive either active AADvac1 or matching placebo.
  Interventions: Biological: AADvac1
- Regimen B: LM11A-31 (Experimental): Participants are randomized to receive either active LM11A-31 or matching placebo.
  Interventions: Drug: LM11A-31

INTERVENTIONS:
Biological: AADvac1 — Active immunotherapy
  Arms: Regimen A: AADvac1
Drug: LM11A-31 — Small molecule
  Arms: Regimen B: LM11A-31

SUMMARY:
The Progressive Supranuclear Palsy Clinical Trial Platform (PTP) is a multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of PSP.

DETAILED DESCRIPTION:
The Progressive Supranuclear Palsy Clinical Trial Platform (PTP) is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial.

In this trial, multiple investigational products for PSP will be tested simultaneously or sequentially. Each investigational product will be tested in a regimen. Each regimen consists of a placebo-controlled trial, meaning that the active investigational product and matching placebo will be tested in each regimen.

The additional details that govern the testing of each investigational product will be summarized in separate regimen-specific appendices (RSAs). Each regimen will have a separate ClinicalTrials.gov posting, which will include specific information about the regimen. All regimen-specific outcome measures will be detailed in each regimen posting.

Participants will have an equal chance to be randomized to all regimens that are active at the time of screening. Once randomized to a regimen, participants will be randomized as outlined for each individual regimen to either study drug or placebo.

New regimens will be continuously added as new investigational products become available. PTP will enroll additional participants as each new regimen becomes available.

PTP is expected to launch with the following regimen:

* Regimen A: AADvac1
* Regimen B: LM11A-31

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of possible or probable PSP Richardson's Syndrome as defined by the 2017 Movement Disorder Society (MDS) criteria.
2. Presence of PSP symptoms for ≤5 years at screening (based on the best judgment of the site PI).
3. Mini-Mental State Examination (MMSE) score at screening of ≥25.
4. Able to walk at least 10 steps with minimal assistance (e.g., one arm for safety, but not postural support).
5. Stable doses of permitted medications as described per protocol for 30 days prior to screening.
6. Resides at home or in the community (assisted living is acceptable).
7. As assessed by the site PI, participant is likely to be able to comply with the protocol for the duration of the study, and has adequate vision, hearing (hearing aid permitted), and literacy (English or Spanish) sufficient for compliance with the required testing procedures.

Exclusion Criteria:

1. Females who are breastfeeding or pregnant (as documented by a urine pregnancy test) during screening, or plan to become pregnant during the study.
2. Females of childbearing potential who did not use a highly effective method of contraception within 28 days of screening and/or are not willing to use a highly effective method of contraception for the duration of their participation in the study.
3. Lacks good venous access such that multiple blood draws would be precluded.
4. Weighs less than 40kg, or more than 136kg at screening.
5. Blood transfusion within 4 weeks of screening.
6. Contraindications to MRI studies, including metal (ferromagnetic) implants, a cardiac pacemaker that is not compatible with MRI, and/or severe claustrophobia.
7. Screening MRI scan showing structural evidence of alternative pathology not consistent with PSP that could explain a substantial portion of the participant's symptoms as indicated by the central MRI read.
8. Any unstable and/or clinically significant medical condition likely to hamper the evaluation of safety and/or efficacy of study drug (e.g., clinically significant reduction in serum B12 or folate levels, clinically significant abnormalities of thyroid function, stroke, or other cerebrovascular or cardiovascular conditions), as per the site PI's judgment.
9. History of severe allergic reaction (e.g., anaphylaxis) including but not limited to: severe allergic reaction to previous vaccines, foods, and/or medications.
10. Hospitalization within 30 days prior to screening or baseline.
11. Infections or major surgical procedures within 3 months prior to screening, judged to be clinically significant by the site PI.
12. Myocardial infarction within 1 year prior to baseline, unstable angina pectoris, symptomatic congestive heart failure.
13. History of cancer within the past 5 years other than treated skin squamous cell carcinoma, basal cell carcinoma, and melanoma in-situ, localized prostate cancer not requiring treatment, or prostate or breast cancer, which have been fully removed and are considered cured.
14. History or presence of immunological or inflammatory conditions, including neurological disorders, meningitis or meningoencephalitis.
15. History or presence of epilepsy requiring ongoing use of antiepileptic medications. Antiepileptic medications are permitted for pain or psychiatric use per the protocol.
16. DSM-5 criteria for drug or alcohol abuse or dependence currently met within the past 5 years.
17. Clinically significant abnormal vital signs including sustained sitting blood pressure >160/100 mm Hg.
18. Diabetes mellitus with hemoglobin A1c (HbA1c) levels of ≥8.0%.
19. Known history of human immunodeficiency virus (HIV-1 or 2).
20. Known history of acute/chronic hepatitis B or C unless treated curatively.

Ages: 41 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression | 52 weeks
  Change in disease severity as measured by the 15-item modified Progressive Supranuclear Palsy Rating Scale (mPSPRS-15) in which the minimum score is 0 and the maximum score is 52, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Disease progression | 52 weeks
  Change in disease severity as measured by the 10-item modified Progressive Supranuclear Palsy Rating Scale (mPSPRS-10) in which the minimum score is 0 and the maximum score is 30, with higher scores indicating a worse outcome.
Disease progression | 52 weeks
  Change in disease severity as measured by the 28-item Progressive Supranuclear Palsy Rating Scale (28-item PSPRS) in which the minimum score is 0 and the maximum score is 100, with higher scores indicating a worse outcome.
Experiences of daily living | 52 weeks
  Change in experiences of daily living over time as measured by the Cortical Basal ganglia Functional Scale (CBFS) in which the minimum score is 0 and the maximum score is 124, with higher scores indicating a worse outcome.
Activities of daily living | 52 weeks
  Change in activities of daily living over time as measured by the Schwab and England Activities of Daily Living Scale (SE-ADL) in which the minimum score is 0% and the maximum score is 100%, with lower scores indicating a worse outcome.
Disease severity | 52 weeks
  Change in disease severity over time as measured by the Clinical Global Impression of disease severity (CGIds) using a 7-point scale, ranging from 1 (normal, not ill) to 7 (extremely ill), with a higher score indicating a worse outcome.
Disease progression | 52 weeks
  Change in disease severity over time as measured by the Clinical Global Impression of Change (CGIC) using a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change.
Health-related quality of life | 52 weeks
  Change in quality of life over time as measured by the EuroQoL 5 Dimension - 5 Level (EQ-5D-5L) questionnaire in which the minimum score is 0 and the maximum score is 1, with lower scores indicating a worse outcome.
Brain volume | 52 weeks
  Change in volume in midbrain, pontine and other regions over time as measured by volumetric MRI.
Neurodegeneration | 52 weeks
  Change in plasma neurofilament light chain (NfL) concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco; Irene Litvan, MD, Principal Investigator — University of California, San Diego; Julio Rojas-Martinez, MD, PhD, Principal Investigator — University of California, San Francisco; Anne-Marie Wills, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol